CLINICAL TRIAL: NCT03135678
Title: Observe Pilot, a Prospective Study to Verify the Feasibility of Collecting a Broad Variety of Individual Health Data
Brief Title: Study to Verify the Feasibility of Collecting a Broad Variety of Individual Health Data
Status: Completed | Type: Observational
Sponsor: Hilbert Paradox NV (Industry)
Responsible Party: Sponsor
Other Study IDs: OBS_001
Record Dates: First submitted 2017-04-22; First posted 2017-05-01 (Actual); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of the OBSERVE PILOT is to verify the feasibility of collecting individual health data which is obtained through blood samples, continuous monitoring devices, medical imaging, a questionnaire, and a blood pressure monitor.

Feasibility of collecting individual health data within the OBSERVE PILOT is described as the ease of gathering a broad variety of data by assessing: (1) the willingness of the subjects to participate in the study, (2) the logistics corresponding with the variety, and (3) the regulatory aspects of gathering a broad variety of data.

ELIGIBILITY:
Inclusion Criteria:

* The subject is able and willing to provide written informed consent prior to research specific data collection.
* The subject must be older than 18 years old.

Exclusion Criteria:

* The subject should not suffer from glaucoma.
* The subject should not be allergic to eye drops.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The population is a healthy population.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2017-05-12 (Actual); Primary Completion 2017-05-23 (Actual); Study Completion 2017-05-23 (Actual)

PRIMARY OUTCOMES:
The number of subjects willing to join the study | Through study completion, an average of 6 months
  The number of subjects invited compared to the number of patients willing to join
The number of health data types that were measured | Through study completion, an average of 6 months
  The number of health data types that were measured compared to the number of health data types anticipated

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Verheye, MD, PhD, Principal Investigator — Director at Hilbert Paradox
Locations (1):
- General Practice, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: No